CLINICAL TRIAL: NCT02275572
Title: Clinical and Economical Assessment of an Intervention to Reduce Potentially Inappropriate Medication in Polymedicated Elderly Patients
Acronym: REMEI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari del Maresme (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 05/12
Record Dates: First submitted 2014-10-21; First posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Polypharmacy; Elderly

ARMS (2):
- Pharmacist Intervention (Experimental): Primary care pharmacist apply the GP-GP algorithm to each drug with the support of STOPP criteria, Beers and / or recommendations CatSalut. The pharmacist submit to doctor his findings and reach a consensus and decide which recommendations will be presented to patient.
  Interventions: Procedure: Pharmacist Intervention
- Control (No Intervention): Usual procedure.

INTERVENTIONS:
Procedure: Pharmacist Intervention
  Arms: Pharmacist Intervention

SUMMARY:
Objective: To evaluate the clinical and economic impact of the application of an algorithm to improve the adequacy and safety of pharmacotherapy in elderly polymedicated (receiving 8 or more medications), not institutionalized.

Design: randomized, open, multicenter and two branches of parallel intervention clinical trial.

Intervention Study: primary care pharmacist apply the GP-GP algorithm to each drug with the support of STOPP criteria, Beers and / or recommendations CatSalut. The pharmacist submit to doctor his findings and reach a consensus and decide which recommendations will be presented to patient. Control intervention: usual procedure.

Main outcome measures: a) Discontinued medications, changed or changing doses, b) GP consultations, hospital emergency department and hospital admissions for acute illness, c) pharmaceutical expenditure, d) restart medication e) complications underlying diseases. Follow-up control at 1 month (security) and at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 70 years or more
* Currently receiving eight or more drugs, except ointments and administered via topical nonprescription
* Give their informed written consent to participate in the study.

Exclusion Criteria:

* Estimated life expectancy less than 6 months.
* Active cancer
* Participation in any other clinical trial or program for evaluation of medication in the elderly.
* Institutionalized in nursing homes.
* Surgical intervention scheduled for the next 6 months

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 503 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with medications discontinued, reduced dose or changed. | baseline, 3, 6 and 12 months
Number of discontinued medications, changed or changing doses. | baseline, 3, 6 and 12 months

SECONDARY OUTCOMES:
Resumption of medication | 3, 6 and 12 months
Medication adherence | baseline, 3 and 6 months
  Morisky-Green questionnaire
Quality of life | baseline, 3 and 6 months
  EuroQoL questionnaire
Pharmaceutical recommendations acceptance rate | baseline
Healthcare resource consumption | 3, 6 and 12 months
  Number of visits to Primary care center, Number of visits to hospital emergency department, Number of hospital admission, Number of outpatients hospital visits.
Mortality | 3, 6 and 12 months

REFERENCES:
- [Derived] Campins L, Serra-Prat M, Gozalo I, Lopez D, Palomera E, Agusti C, Cabre M; REMEI Group. Randomized controlled trial of an intervention to improve drug appropriateness in community-dwelling polymedicated elderly people. Fam Pract. 2017 Feb;34(1):36-42. doi: 10.1093/fampra/cmw073. Epub 2016 Sep 7. PMID 27605543